CLINICAL TRIAL: NCT04664062
Title: Comparing Home, Office, and Telehealth Induction for Medication Assisted Treatment for Opioid Use Disorder
Acronym: HOMER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Academy of Family Physicians National Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-1692
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Opioid-use Disorder; Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Opiate Substitution Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home (Active Comparator): This induction arm is asynchronous and unobserved. The home induction is done primarily by the participant in their home or current residence. The participant receives instruction on induction process from clinic team at an in-person or telehealth visit. Home induction is initiated by the participant at a time and place (other than the practice) determined by the participant. The participant determines when to stop taking opioids, begins withdrawal, monitors symptoms, administers the SOWS, and determines when to take first dose of medication, per the instructions and protocol provided. The clinic team does not observe or have contact with the participant while the participant undergoes these steps or takes the first dose. The participant continues this process for additional doses. Follow-up contact with clinic team may occur after the first or second day, typically within a week.
  Interventions: Behavioral: Medication Assisted Treatment
- Office (Active Comparator): This induction arm is synchronous and observed by the clinical team. The participant receives instruction from clinic team at an in-person or telehealth visit. On a pre-determined day, the participant stops taking opioids and comes to office with mild to moderate withdrawal. The clinic team monitors the participant, assesses symptoms, administers COWS to determine time of first dose of medication, and administers first dose with the participant. The clinic team observes and has in-person contact with the participant. Office induction includes the observed administration of the first dose, followed by observation and evaluation 30-60 minutes after the first dose. After 30-60 minutes of observation, the clinic team and participant decide whether to administer the second dose in the office or for the participant to leave the clinic to administer subsequent doses. On rare occasions, a second dose may not be needed (if the participant has a low COWS score after just one dose).
  Interventions: Behavioral: Medication Assisted Treatment
- Telehealth (Active Comparator): This induction arm is synchronous via phone or video contact and observed. The participant receives instruction on induction process from clinic team at an in-person or telehealth visit. The participant undergoes the same process as an office induction but from a location other than the clinic. Like an office induction, the participant has regular contact with someone from the practice team on Day 1 of induction. Prior to initiating the first dose, the participant has contact by phone or video with the clinic team to assess symptoms and determine level of withdrawal (using COWS or SOWS). The administration of the first dose of medication is determine by the clinic team during phone or video contact, and the clinic team is in contact with the participant by phone or video when the first dose is taken. This process continues through the second and possible third dose. The participant is re-assessed via video or phone regularly by clinic staff and prescriber throughout this process.
  Interventions: Behavioral: Medication Assisted Treatment

INTERVENTIONS:
Behavioral: Medication Assisted Treatment — All subjects will undergo MAT induction with buprenorphine. Participants will be randomized to the behavioral aspects of induction, specifically comparing office induction vs home vs synchronous telehealth induction.

SUMMARY:
HOMER is a national study comparing three methods of induction for Medication Assisted Treatment (MAT) for Opioid Use Disorder (OUD); home versus office versus telehealth-based inductions. This study will help determine if certain patient and practice characteristics make patients better candidates for one method over the others. Results will help fill a gap in the evidence around effectively treating OUD with MAT in primary care settings.

DETAILED DESCRIPTION:
Office-based Opioid Treatment (OBOT) is the primary care or ambulatory care provision of medication assisted treatment (MAT) for patients suffering opioid use disorder (OUD). MAT with buprenorphine in primary care clinics is a proven strategy to treat opioid use disorder (OUD) and is slowly becoming accessible to patients through primary care. Treating patients with buprenorphine involves an initial induction, during which patients discontinue their opioids, begin withdrawal, and receive the first few doses of buprenorphine. National guidelines for OBOT have focused on observed, office-based induction to begin MAT. Over the years, unobserved, home MAT inductions have also been used and shown to be safe and effective. Individually, each induction strategy is evidence-based, guideline concordant care. In light of the current COVID-19 pandemic, inductions are also being conducted via telehealth using synchronous audio or video observation. Most research, on which the current guidelines are based, examined short-term outcomes. However, OUD is a chronic condition. MAT often involves intermittent return to illicit opioid use and treatment lapses, resulting in multiple attempts to remain in long-term treatment. Important differences between the activities that occur during home, office-based, and telehealth induction might influence short-term stabilization, long-term maintenance treatment, and quality of life outcomes. No large-scale, multi-center, randomized comparative effectiveness research has compared induction method on long-term outcomes for patients suffering from OUD seen in primary care settings.There is currently insufficient evidence to recommend home induction (asynchronous, unobserved), office induction (synchronous, observed), or telehealth induction (synchronous phone or video contact, observed).

Acknowledging the dire need for increased access to effective treatment for OUD, patients and providers are eager to better understand if home, office-based, or telehealth induction in the primary care setting leads to more successful short-term stabilization and long-term maintenance treatment and patient outcomes. They also question whether certain patient characteristics, such as substance use history, executive function, and social determinants of health, are associated with better long-term outcomes in patients receiving one method versus the others. We propose a comparative effectiveness research study, randomized at the patient level, to compare short-term stabilization and long-term maintenance treatment outcomes of home induction (asynchronous, unobserved), office induction (synchronous, observed), or telehealth induction (synchronous phone or video contact, observed) for patients suffering from OUD and opioid dependence.

ELIGIBILITY:
Inclusion Criteria:

Ages 16 and older Identified by their clinician as having opioid dependence and either 1) addiction as defined by DSM-V criteria for OUD and/or 2) chronic pain with long-term, high dose opioid use (greater than one year and morphine equivalent daily dose higher than recommended by the CDC).

Seeking or agreeing to receive medication assisted treatment (MAT) with buprenorphine or Suboxone (buprenorphine/naloxone).

Agree to be randomly assigned to undergo MAT induction with one of the three methods being compared in this study.

* home induction (asynchronous, unobserved)
* office induction (synchronous, observed)
* telehealth induction (synchronous phone or video contact, observed) Agree to answer a set of survey questions four times over a nine month period (at the time of enrollment plus 1, 3, and 9 months after starting treatment.

Exclusion Criteria:

Hypersensitivity to buprenorphine or naloxone. Are known to have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels greater than five times normal.

Are diagnosed with severe, untreated psychiatric illness. Have a preference for one of the MAT induction methods and do not want to be randomly assigned to one.

Ages: 16 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of days patient took buprenorphine | 270 days
  Determined by prescription refills and patient self-report of number of days buprenorphine taken.
Number of days patient took illicit opioids | 270 days
  Determined by a patient self-report of the number of days they took other opioids and urine opioid test results.
Took buprenorphine on >80% of days | 270 days
  Determined by initial prescription and refills, a patient self-report of number of days buprenorphine taken, and urine buprenorphine results.
Percent (%) of patients that took other opioids on <10% of days | 270 days
  Determined by a patient self-report of the numer of days they took other opioids and urine opioid test results.

SECONDARY OUTCOMES:
Social Determinant of Health and Quality of Life | 270 days
  Patient surveys completed per clinical care on quality of life (e.g., symptoms, side effects, depression), social connectedness, loneliness, and other select determinants of health.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado, Denver, Colorado
  - American Academy of Family Physicians National Research Network, Leawood, Kansas

IPD SHARING:
Plan to Share IPD: No